CLINICAL TRIAL: NCT01071499
Title: Pharmacokinetics of Oral Morphine and Pharmacogenomics of CYP2D6 and UGT2B7, in an Urban Pediatric Population (2 - 6 Years of Age) Presenting for Elective Surgery
Brief Title: Pharmacokinetics of Oral Morphine and Pharmacogenomics of CYP2D6 and UGT2B7, in an Urban Pediatric Population Presenting for Elective Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Carolyne Montgomery, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H09-03286
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: pharmacokinetics; pharmacogenetics; morphine; children
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Subjects recruited will be block assigned to one of the three doses of morphine. Sampling will be done for 4 hrs to determine the key pharmacokinetic parameters.
  Interventions: Drug: Morphine
- 2 (Active Comparator): Subjects recruited will be block assigned to one of the three doses of morphine. Sampling will be done for 4 hrs to determine the key pharmacokinetic parameters.
  Interventions: Drug: Morphine
- 3 (Active Comparator): Subjects recruited will be block assigned to one of the three doses of morphine. Sampling will be done for 4 hrs to determine the key pharmacokinetic parameters.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — One dose of morphine (0.1 mg/kg)
  Arms: 1
Drug: Morphine — One dose of morphine (0.2 mg/kg)
  Arms: 2
Drug: Morphine — One dose of morphine (0.3 mg/kg)
  Arms: 3

SUMMARY:
The purpose of this study is to identify and collect samples from children who have taken a single oral dose of the pain medication morphine, and to determine the genetic differences in the way children metabolize (break down in the body and how it affects them) morphine.

DETAILED DESCRIPTION:
Hypothesis:

Oral morphine will produce more reliable peak plasma morphine concentrations and more reliable analgesia than codeine, which is currently the drug of choice.

Background:

Codeine is the most commonly used oral opiate for analgesia in children. Codeine is a pro-drug that requires activation by the isozyme CYP2D6. Genetically determined variations in the activity of CYP2D6 can result in inappropriately low analgesic efficacy due to inadequate conversion of the drug in "poor-metabolizers" and conversely, adverse reactions such as respiratory depression and death in "ultra-metabolizers". In some ethnic groups as many as 40% of patients may be susceptible to concentration-dependent toxicity from greater than expected metabolism of codeine to morphine. We hypothesize that oral morphine is a feasible and safe alternative to codeine. The primary aim of this study is to define and trial an appropriate dose of morphine to provide children with effective and reliable perioperative analgesia with a minimum risk of adverse drug effects. A secondary aim is to investigate the pharmacogenetics of codeine and morphine metabolism in children.

Specific Objectives:

The pharmacokinetic properties of 3 (0.1 mg/kg, 0.2 mg/kg or 0.3 mg/kg) doses of oral morphine will be described. We will determine the dose of oral morphine that results in a peak plasma concentration that occurs within 60 - 90 min and results in the analgesic therapeutic range (10 - 40 ng/mL). Pharmacogenetic profiles for two key enzymes involved in codeine and morphine metabolism (CYP2D6 and UGT2B7) will be determined.

Methods:

After obtaining institutional review board approval, and written parental informed consent, we will recruit 45 children for Phase I aged 2-6 years undergoing elective surgery. A perceived ethnicity questionnaire will also be administered. Subjects recruited for Phase I will be block assigned to one of the three doses of morphine. In Phase I, sampling will be done for 4 hrs to determine the key pharmacokinetic parameters including Tmax, Cmax and AUC. Monitoring will occur throughout and analgesic efficacy and adverse effects will be measured post-operatively. All subjects will receive 24 hr telephone follow up for analgesic efficacy and adverse drug effects.

Data Analysis: All continuous parametric data (weight, age, BMI) will be analyzed using t-tests. Non-parametric ordinal data such as pain scores will be analyzed by the Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* 2 - 6 years of age
* ASA 1 & 2 elective surgical patients - Procedures requiring opioid analgesia - Minimal hospital stay of 4 hrs
* Informed consent

Exclusion Criteria:

* Allergy or adverse reaction to morphine
* Contraindication to morphine analgesia, such as a potential difficult airway -- Abnormal hepatic or renal function known by history or available laboratory results
* Current regular opioid use
* Surgical or anesthetic contraindication to oral premedication such as gastro-esophageal reflux disease
* Children with a BMI of <10'ile or >90'ile
* Declines study participation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
1 mL blood sample will be obtained at 30, 60, 90, 120, 180 and 240 min after morphine administration. | 4 hours

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability (FLACC) pain score | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Carolyne Montgomery, Dr., Principal Investigator — University of British Columbia; Gillian Lauder, Dr., Study Director — University of British Columbia; Katherine Brand, Dr., Study Director — University of British Columbia; Bruce Carleton, Dr., Study Director — University of British Columbia; Gideon Koren, Dr., Study Director — University of British Columbia; Michael Rider, Dr., Study Director — University of British Columbia
Locations (1):
- British Columbia Children's Hospital-Dept of Anesthesia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Velez de Mendizabal N, Jimenez-Mendez R, Cooke E, Montgomery CJ, Dawes J, Rieder MJ, Aleksa K, Koren G, Jacobo-Cabral CO, Gonzalez-Ramirez R, Castaneda-Hernandez G, Carleton BC. A Compartmental Analysis for Morphine and Its Metabolites in Young Children After a Single Oral Dose. Clin Pharmacokinet. 2015 Oct;54(10):1083-90. doi: 10.1007/s40262-015-0256-4. PMID 25773480